CLINICAL TRIAL: NCT03513640
Title: Prospective Cohort for Finding Risk Factors of Meconium Obstruction and Respiratory Distress Syndrome in Preterm Infants
Brief Title: Risk Factors of Meconium Obstruction and Respiratory Distress Syndrome in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ee-Kyung Kim, Professor, Seoul National University Hospital
Other Study IDs: 1705-073-853
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Meconium Obstruction of Prematurity; Respiratory Distress Syndrome in Premature Infant
MeSH Terms: conditions — Meconium Ileus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample at birth for citrulline level analysis urine sample at the first day of life for fatty acid binding protein analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although the pathophysiology of meconium obstruction of prematurity (MOP) is not clear, it is known that the decrease of the intestinal peristalsis due to decreased intestinal perfusion during antenatal or perinatal period. Recently, the level of citrulline has been used as an index of function and injury of the small intestine State. This study aimed to evaluate citrulline level of cord blood as a marker for early detection and observe changes in intestinal blood flow in MOP patient.

And We aimed to confirm the efficacy of the AT/ET ratio (ratio of the pulmonary artery time-to-peak velocity interval to the right ventricular ejection time) of the prenatal pulmonary artery as a noninvasive predictor of neonatal respiratory distress syndrome.

ELIGIBILITY:
Inclusion Criteria:

* premature infants born less than 34 weeks from mother with pregnancy induced hypertension, pre-eclampsia or eclampsia

Exclusion Criteria:

* major congenital anomalies
* infants with hypotension while using inotropics

Max Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants born less than 34 weeks who were admitted in neonatal intensive care unit at Seoul National University Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of citrulline level between the meconium obstruction group and the normal feeding advance group | within 6 hours after birth
  check the citrulline llevel from blood at birth
Comparison of prenatal AT/ET ratio of fetal pulmonary artery between respiratory distress syndrome group and the normal respiration group | within 10 days before delivery
  Check the AT/ET ratio of fetal pulmonary artery within 10 days before birth

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes